CLINICAL TRIAL: NCT06989892
Title: Comparing Super High-flux and High-flux Dialyzer Performance Among Hemodialysis Patient With Sepsis : a Randomized Control Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Navamindradhiraj University (Other)
Responsible Party: Principal Investigator, Punnawit Laungchuaychok, Dr., Navamindradhiraj University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 205/66
Record Dates: First submitted 2024-07-24; First posted 2025-05-25 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: The Efficacy and Safety for Super High-flux Dialyzer in Case of Sepsis in ESKD; End Stage Kidney Disease (ESRD); Sepsis
Keywords: Superhighflux; hemodialysis; end stage kidney disease; sepsis
MeSH Terms: conditions — Kidney Failure, Chronic; Sepsis

STUDY DESIGN:
Intervention Model Description: Comparing the mortality in sepsis condition between two groups of ESKD patient who underwent hemodialysis with superhighflux and highflux dialyzer
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ESKD patient with sepsis who dialyzed with super high flux (Experimental): Patients received dialysis with Superhigh-flux dialyzer
  Interventions: Device: Super High-flux dialyzer (Elisio 19HDx)
- ESKD with sepsis who dialyzed with high flux dialyzer (Active Comparator): Patients received dialysis with High-flux dialyzer
  Interventions: Device: High-flux dialyzer (Elisio 19H)

INTERVENTIONS:
Device: Super High-flux dialyzer (Elisio 19HDx) — Dialysis with Super High-flux dialyzer for intervention group
  Arms: ESKD patient with sepsis who dialyzed with super high flux
Device: High-flux dialyzer (Elisio 19H) — Dialysis with High-flux dialyzer for control group
  Arms: ESKD with sepsis who dialyzed with high flux dialyzer

SUMMARY:
Comparing the efficacy of superhigh-flux dialyzer with high-flux dialyzer in ESKD patient who have sepsis to improve mortality and sepsis outcome, an open label randomized control trial.

DETAILED DESCRIPTION:
Sepsis in people who have ESKD is the risk of developing poor outcome. Cytokines play a role in the process of sepsis and cause the worsening clinical outcome despite definitive antibiotic treatment. Superhigh-flux dialyzer has a larger molecular weight cut off (MWCO) clearance, include cytokine, could contribute to improved sepsis management in individuals with ESKD. This study is conducted to prove the efficacy of super high-flux dialyzer comparing with high-flux dialyzer in case of mortality reduction for regular hemodialysis ESKD patients.

Method This study is an open label single center randomized control trial. We randomized ESKD patients who have sepsis condition with high interleukin-6 (IL-6 > 50 pg/ml).

The participants were allocated to super high-flux dialyzer group and high flux dialyzer group, stratified with diabetes, vascular access, and septic shock.

We excluded; patient who needed dialysis with continuous kidney replacement therapy, vulnerable patient, include pregnant woman, patient who closed and patient who expected to pass away within the 24 hours. We aim to enroll total 202 participants; divided equally in each arm. According to our protocol, non reused super high-flux dialyzer and high-flux dialyzer are used in the same assigned patient in first week without crossing over. The standard of care of sepsis and antibiotic are provided in both groups without intervening of researcher and our protocol. The primary endpoint is 28 days of mortality. The secondary outcome include cardiovascular death, rate reduction of IL-6 after dialysis, days of hospitalization, ventilator free days and complication of dialysis are also monitored.

ELIGIBILITY:
Inclusion Criteria:

* ESKD patients who have sepsis condition with high interleukin-6 (IL-6 > 50 pg/ml)

Exclusion Criteria:

* Patients who needed dialysis with continuous kidney replacement therapy, vulnerable patient, include pregnant woman, patient who expected to pass away within the 24 hours.
* Patients who have the history of allergic dialyzer reaction to dialyzer which used in this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Estimated)
Dates: Start 2024-07-25 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Comparing the reduction of all cause death at 28 days | 28 days
  Comparing the efficacy to reduce all cause death at 28 days between Super High-flux dialyzer with High-flux dialyzer in ESKD with sepsis

SECONDARY OUTCOMES:
Comparing the difference of blood level of IL-6, ESR, CRP and albumin, before and after of the first dialysis session, in each group. | 7 days
The duration of inotrope weaning | 14 days
The duration of hospitalization | 28 days
Ventilator free days | 28 days
The incidence of intradialytic hypotension | 28 days
The incidence rate of complication of dialyzer in each group | 28 days
  The incidence rate of complication of dialyzer; allergic reaction, clotting of dialyzer etc.
The adequacy profile of dialysis in both groups | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Punnawit Laungchuaychok, MD, Principal Investigator — Navamindradhiraj University; Wanjak Pongsittisak, MD, Study Chair — Navamindradhiraj University
Locations (1):
- Navamindhradhiraj university, Dusit, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zhou F, Peng Z, Murugan R, Kellum JA. Blood purification and mortality in sepsis: a meta-analysis of randomized trials. Crit Care Med. 2013 Sep;41(9):2209-20. doi: 10.1097/CCM.0b013e31828cf412. PMID 23860248
- [Background] Gharamti AA, Samara O, Monzon A, Montalbano G, Scherger S, DeSanto K, Chastain DB, Sillau S, Montoya JG, Franco-Paredes C, Henao-Martinez AF, Shapiro L. Proinflammatory cytokines levels in sepsis and healthy volunteers, and tumor necrosis factor-alpha associated sepsis mortality: A systematic review and meta-analysis. Cytokine. 2022 Oct;158:156006. doi: 10.1016/j.cyto.2022.156006. Epub 2022 Aug 28. PMID 36044827
- [Background] Sarnak MJ, Jaber BL. Mortality caused by sepsis in patients with end-stage renal disease compared with the general population. Kidney Int. 2000 Oct;58(4):1758-64. doi: 10.1111/j.1523-1755.2000.00337.x. PMID 11012910
- [Background] Song J, Park DW, Moon S, Cho HJ, Park JH, Seok H, Choi WS. Diagnostic and prognostic value of interleukin-6, pentraxin 3, and procalcitonin levels among sepsis and septic shock patients: a prospective controlled study according to the Sepsis-3 definitions. BMC Infect Dis. 2019 Nov 12;19(1):968. doi: 10.1186/s12879-019-4618-7. PMID 31718563
- [Background] Abe M, Masakane I, Wada A, Nakai S, Nitta K, Nakamoto H. Super high-flux membrane dialyzers improve mortality in patients on hemodialysis: a 3-year nationwide cohort study. Clin Kidney J. 2021 Sep 28;15(3):473-483. doi: 10.1093/ckj/sfab177. eCollection 2022 Mar. PMID 35211304
- [Background] Pongsittisak W, Satpanich P, Jaturapisanukul S, Keawvichit R, Prommool S, Trakranvanich T, Ngamvichukorn T, Kurathong S. Medium Cut-Off versus Low-Flux Dialyzers in Hemodialysis Patients with COVID-19: Clinical Outcomes and Reduction in Interleukin-6. Blood Purif. 2023;52(6):591-599. doi: 10.1159/000530162. Epub 2023 May 5. PMID 37231799
- See also: Related Info — https://drive.google.com/drive/folders/10hokBrbRQS5F9rYjx2JK4JZaBuIOVHqS